CLINICAL TRIAL: NCT05240560
Title: A Multisite Randomized Clinical Trial Evaluating Efficacy and Safety of BP1.3656 vs Placebo in Patients With Fatigue Following Ischemic Stroke
Brief Title: Proof of Concept Study Evaluating BP1.3656 in Patients With Fatigue Following Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P20-04 / BP1.3656; 2020-006006-23 (EudraCT Number)
Record Dates: First submitted 2022-01-20; First posted 2022-02-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fatigue
Keywords: Post-stroke fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo tablets will be identical in appearance to the BP1.3656 tablets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP1.3656 (Experimental): 1 tablet of 30 microgram (µg), 60µg or 90µg of BP1.3656 per day
  Interventions: Drug: BP1.3656
- Placebo (Placebo Comparator): 1 tablet of matching placebo per day
  Interventions: Drug: BP1.3656

INTERVENTIONS:
Drug: BP1.3656 — Histamine H3 receptor antagonist/inverse agonist

SUMMARY:
Multicenter, randomized, double blind, parallel-group, placebo-controlled proof of concept study evaluating efficacy and safety of BP1.3656 in patients with fatigue following ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years old or more;
* Diagnosis of ischemic stroke at least one month and not more than six months prior to screening;
* Persistent fatigue since the stroke with a score ≥ 50 across all domains of the Multidimensional Fatigue Inventory (MFI-20);
* Modified Rankin Score (mRS) < 3;
* Capability to participate in all study tests according to the investigator;
* Patient must voluntarily express a willingness to participate in this study, sign and date an informed consent prior to any study specific procedure;
* Females of child-bearing potential must have a negative pregnancy test performed at the screening and randomization visits and use a medically accepted effective method of birth control, agree to continue this method for the duration of the study up until three weeks after last treatment intake.

Exclusion Criteria:

* Any identified etiology for fatigue other than stroke (except post-stroke depression) according to the investigator;
* History of psychosis;
* Current severe psychiatric disorder, e.g. schizophrenia, bipolar disorder, severe depression, or organic brain syndrome preventing the patients from completing study assessments;
* Patients at risk of suicide according to the investigator;
* Major cognitive disorders, dementia according to the investigator;
* History of epilepsy or seizures disorder;
* History of alcohol or drugs (i.e. cannabis, cocaine, amphetamines or opioids) (ab)use/dependence within the 12 months prior to screening or with a positive drug test at screening;
* Glomerular filtration rate <60 mL/min/1.73m² according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula;
* Clinically significant cardiovascular abnormalities (including clinically relevant ECG abnormalities) or, clinically significant hematological, neurological, endocrine abnormalities, severe hepatic impairment or Liver Function Tests (ASAT, ALAT) > 3 ULN, or abnormal clinical laboratory results (in most cases > 3ULN);
* Other active clinically significant illness, infection, acid-related gastric disorder, or neoplastic pathology within the last 3 years (patients with fully cured non-melanoma skin cancer or in-situ carcinoma of the cervix are eligible) which could interfere with the study conduct or counter-indicate the study treatments or place the patient at risk during the trial or compromise his/her study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI-20) global score | Week 8
  20-item self-report instrument designed to measure fatigue experienced by the participant lately scored from 20 to 100. Higher scores show higher levels of fatigue.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) as assessed by AEs collection | Week 8
  Safety assessment of BP1.3656 based on adverse events (AEs) reporting during treatment period.
Change in Systolic blood pressure (BP) measurement | From baseline to Week 8
  Safety assessment of BP1.3656 based on the measurement of systolic blood pressure in units of millimeters of mercury (mmHg)
Change in Diastolic blood pressure (BP) measurement | From baseline to Week 8
  Safety assessment of BP1.3656 based on the measurement of Diastolic blood pressure in units of millimeters of mercury (mmHg)
Change in pulse | From baseline to Week 8
  Safety assessment of BP1.3656 based on the measurement of pulse in beats/minute

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassetti, MD, Prof., Principal Investigator — Inselspital Bern, Department of Neurology, Bern, Switzerland
Locations (2):
- Hôpital Pellegrin - CHU BORDEAUX, Bordeaux, France
- Inselspital Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No